CLINICAL TRIAL: NCT02759159
Title: The Study of Brain Functional Network Modulatory Mechanism of Alzheimer's Disease Using Acupuncture at the "Four-gate" Acupoints
Brief Title: The Study of Mechanism of Alzheimer's Disease Using Acupuncture Based on fMRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, likuncheng, Head of Radiology Department, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 81471649
Record Dates: First submitted 2016-04-14; First posted 2016-05-03 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AD-true acupuncture (Experimental): True acupuncture at the "four-gate"acupoints will be administered on AD patients
  Interventions: Procedure: true acupuncture
- AD-sham acupuncture (Sham Comparator): Sham acupuncture at the "four-gate"acupoints will be administered on AD patients
  Interventions: Procedure: sham acupuncture
- Mild Cognitive Impairment(MCI)-true acupuncture (Experimental): True acupuncture at the "four-gate"acupoints will be administered on MCI patients
  Interventions: Procedure: true acupuncture
- MCI-sham acupuncture (Sham Comparator): Sham acupuncture at the "four-gate"acupoints will be administered on MCI patients
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: true acupuncture — acupuncture at the "four-gate"acupoints, three times per week and last for 6 months
  Arms: AD-true acupuncture; Mild Cognitive Impairment(MCI)-true acupuncture
Procedure: sham acupuncture — acupuncture at the places 1cm from the true "four-gate "acupoints,three times per week and last for 6 months
  Arms: AD-sham acupuncture; MCI-sham acupuncture

SUMMARY:
Alzheimer's disease (AD) is one of the major brain diseases which received more attention in recent years. The disconnection syndrome is the main pathophysiological mechanism leading to cognitive decline in AD patients. Both animal experiment and clinical observation have demonstrated that acupuncture can generate treatment effect on AD patients by moderating the neural pathway directly. However, the underlying mechanism remains unclear. By using resting state functional magnetic resonance imaging (fMRI) method, as well as acupuncture and neurology sciences, investigators will explore the multi-modality data analysis; compare brain connectivity and network parameters changes between pre- and post- acupuncture treatment; analyze the correlation between fMRI changes and neuropsychology test. The present study aims to elucidate the neural mechanism of acupuncture therapy on early AD, provide theoretical evidence from the perspective of functional connectivity.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Alzheimer's Disease Clinical diagnosis of MCI due to Alzheimer's Disease Drug therapy regularly

Exclusion Criteria:

Frontotemporal dementia Lewy body dementia Vascular dementia Severe depression Brain vascular disease Metabolic disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
brain functional connectivity | with in first week after the whole acupuncture treatment
  GE750 3.0T gradient-echo single-shot echo plannar imaging TR=2000ms TE=30ms slice=36 slice thickness=3mm gap=1mm volumes=180

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xuanwu hospital, Beijing, Beijing Municipality
  - Dongfang Hospital,Beijing University of Chinese Medicine, Beijing, Beijing Municipality